CLINICAL TRIAL: NCT05831618
Title: New Rehabilitation Protocol for Patients With Persistent Postural Perceptual Dizziness
Brief Title: New Rehabilitation Protocol for Patients With PPPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Iole Indovina (Unknown)
Responsible Party: Principal Investigator, Marco Tramontano, Head of Rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSL/CE/2024_021
Record Dates: First submitted 2023-03-06; First posted 2023-04-26 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Rehabilitation; Balance; Vestibular Disorder; Dizziness
MeSH Terms: conditions — Vestibular Diseases; Dizziness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Visuo-Vestibular training (Experimental): Interactive Visuo-Vestibular training consists of exercises that stimulate saccadic movements during motor activities on the treadmill. Furthermore, a dynamic blindfolded training will be performed with the support and supervision of the physiotherapist.
  Patients will perform 5 sessions, 1 session per week.
  Interventions: Other: Interactive Visuo-Vestibular training
- Vestibular rehabilitation training (Active Comparator): The conventional vestibular rehabilitation training will train the vestibular reflexes.
  Patients will perform 5 sessions, 1 session per week.
  Interventions: Other: Vestibular rehabilitation training

INTERVENTIONS:
Other: Interactive Visuo-Vestibular training — Dynamic motor activitites aimed to enhance the visuo-vestibular interaction and the sensorial reweighting will be performed for the Interactive Visuo-Vestibular training group.
  Arms: Interactive Visuo-Vestibular training
Other: Vestibular rehabilitation training — Dynamic motor activitites aimed to enhance vestibular reflexes will be performed for the vestibular rehabilitation group
  Arms: Vestibular rehabilitation training

SUMMARY:
The investigators will test a new rehabilitation protocol on patients with persistent postural perceptual dizziness (PPPD). The investigators hypothesize that patients with PPPD, in the absence of vestibular deficits, do not benefit from standard vestibular rehabilitation but instead need a rehabilitation that acts on visual and postural stability, through training of saccadic movements in dynamic contexts of cognitive-motor dual-task and rehabilitation of postural stability.

DETAILED DESCRIPTION:
Persistent postural-perceptual dizziness (PPPD) is a chronic functional vestibular disorder that manifests as a sensation of non-vertiginous dizziness and instability.

The most common triggers of PPPD are peripheral vestibular conditions such as vestibular neuritis (VN) and benign paroxysmal positional vertigo (BPPV), although vestibular migraine, central vestibular disorders and non-vestibular conditions such as panic attacks, minor injuries traumatic brain injury and also orthostatic intolerance have been reported as precipitants of PPPD. PPPD persists after the triggering events have resolved.

The diagnostic criteria for PPPD were established by the Barany Society. Once the negativity of the routine vestibular tests has been ascertained, the diagnosis is based on additional criteria such as the persistence of the symptom of dizziness for most of the time for at least 3 months, the worsening of the symptoms when standing, during active movement or passive, during exposure to moving visual stimulation or to visual stimuli with complex textures.

Existing treatments (e.g., selective serotonin reuptake inhibitors, vestibular habituation) are only partially successful in PPPD.

Methods. Experimental design. Single-blind randomized controlled trial. 40 individuals affected by PPPD will be recruited.

The patients will be randomly divided into 2 groups and evaluated before the rehabilitation training (T0), immediately after the end of the training (T1), 4 weeks after the end of the training (T2) and 8 weeks after the end of the training (T3). All patients will undergo 5 rehabilitation sessions supervised by a physiotherapist with experience in rehabilitation of balance disorders. The experimental group will carry out a interactive visuo-vestibular training (IVV) in order to facilitate postural visual stability and the control group will carry out a conventional vestibular rehabilitation training aimed at training the vestibular reflexes.

The rehabilitation protocols (IVV and vestibular) will consist of 1 session of 40 minutes per week, for a total of 5 sessions.

IVV training consists of exercises that stimulate saccadic movements during motor activities on the treadmill and walking on the treadmill blindfolded with the support and supervision of the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria established for PPPD by the Barany Society (Staab et al., 2017) will be adopted

Exclusion Criteria:

* Patients with neurological, otological or psychiatric disorders other than PPPD will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Dizziness Handicap Inventory (DHI) score | pre-training (T0), immediately after the end of the training (T1), 4 weeks after the end of the training (T2) and 8 weeks after the end of the training (T3)
  DHI.Questionnaire on the severity of dizziness (Dizziness Handicap Inventory, DHI).
  Scores range from 0 to 50; higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes of locomotion parameter linear acceleration measured through wearable inertial sensors | pre-training (T0), immediately after the end of the training (T1), 4 weeks after the end of the training (T2) and 8 weeks after the end of the training (T3)
  Five wireless wearable inertial sensors will be used. Each inertial sensor measures linear accelerations (m/s^2) along its three axes.
  (L4-L5) of the wrists and shins. During 4 specific tasks, the accelerations of the body segments of interest will be measured.
  The motor tasks will be the following:
  1. the 10 Meter Walk Test, a test commonly used to measure walking speed in which the patient is asked to walk 3 times at preferred speed along a 10-metre path;
  2. the Fukuda Stepping Test.
  3. the walk following a path in the shape of an 8, drawn on the floor and with a diameter of each circle of 1.66 m.
Changes of locomotion parameter angular velocities measured through wearable inertial sensors | pre-training (T0), immediately after the end of the training (T1), 4 weeks after the end of the training (T2) and 8 weeks after the end of the training (T3)
  Five wireless wearable inertial sensors will be used. A triaxial gyroscope will measure angular velocities (rad/s) around three axes.
  (L4-L5) of the wrists and shins. During 4 specific tasks, angular velocities of the body segments of interest will be measured.
  The motor tasks will be the following:
  1. the 10 Meter Walk Test, a test commonly used to measure walking speed in which the patient is asked to walk 3 times at preferred speed along a 10-metre path;
  2. the Fukuda Stepping Test.
  3. the walk following a path in the shape of an 8, drawn on the floor and with a diameter of each circle of 1.66 m.
Changes in visual dependence through rod and the disc test | pre-training (T0), immediately after the end of the training (T1), 4 weeks after the end of the training (T2) and 8 weeks after the end of the training (T3)
  Rod and Disk test. In a darkened room (to eliminate external visual cues), participants will be presented with a visual stimulus on a computer monitor consisting of a bar in the center of a disk and a background of rotating disks. Participants will have to align the bar to the Earth vertical, using the arrows on the computer keyboard. Angular realignment errors with respect to the Earth vertical will be measured.
Changes in postural oscillations | pre-training (T0), immediately after the end of the training (T1), 4 weeks after the end of the training (T2) and 8 weeks after the end of the training (T3)
  Measurement of postural oscillations. Through the "Sway" application (https://www.swaymedical.com/), installed on a mobile phone held on the chest with the patient's arms folded, we will measure the personal accelerations related to the maintenance and loss of balance during standard tasks of the mCTSIB (modified clinical test of sensory interaction on balance) and mBESS (modified balance error scoring system) protocols which alternate feet aligned, leg raised, eyes closed or open, stable or foam support.

IPD SHARING:
Plan to Share IPD: No